CLINICAL TRIAL: NCT07025109
Title: Adaptation and Pilot Testing a Behavioral Physical Activity Intervention With Peer Support for Women With HIV and Co-Occurring Hypertension
Brief Title: Assessing Peer Support for Physical Activity in Women With HIV and Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kaylee Crockett, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 300008025; K23HL156758 (NIH)
Record Dates: First submitted 2025-05-30; First posted 2025-06-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: HIV; Hypertension
Keywords: Women; HIV; Hypertension; Physical Activity; Behavioral clinical trial
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer support arm (Experimental): Women in the peer support arm will receive weekly peer contacts via phone or text message to assess progress towards study-assigned physical activity goal/prescription and to provide motivational counseling and support.
  Interventions: Behavioral: Peer support; Behavioral: Exercise Prescription; Behavioral: Blood pressure self monitoring
- Control arm (Active Comparator): Women in the control arm will receive physical activity prescription and home blood pressure monitoring, but will not receive peer support calls.
  Interventions: Behavioral: Exercise Prescription; Behavioral: Blood pressure self monitoring

INTERVENTIONS:
Behavioral: Peer support — Peer support counseling will include phone or text communication to assess goal progress, provide motivational counseling as needed, and to provide social support.
  Arms: Peer support arm
Behavioral: Exercise Prescription — Women will be provided with an exercise prescription (Frequency, Intensity, Time, Type) which may be adjusted weekly for 6 weeks to goal of 150min/week of moderate to vigorous physical activity.
Behavioral: Blood pressure self monitoring — Women will receive a home blood pressure monitor and encourage to record their readings in a log.

SUMMARY:
This clinical trial will assess the acceptability and feasibility of a peer-supported behavioral physical activity intervention for women living with HIV and Hypertension.

DETAILED DESCRIPTION:
An individually randomized pilot trial (N=50) of an adapted behavioral physical activity (PA) intervention will be used to assess the feasibility and acceptability of providing exercise prescription, peer support, and home blood pressure monitoring to women ages 40+ living with HIV and Hypertension. Secondary outcomes to be assessed include systolic and diastolic blood pressure, PA time and intensity, PA self-efficacy, perceived social support, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* woman living with HIV
* age 40 and above
* diagnosed with HTN
* access to a personal phone for study-related phone calls
* willing to wear an accelerometer on their waist or hip for 7 days at beginning and end of 12-week intervention
* able to ambulate independently
* English speaking

Exclusion Criteria:

* Pregnant
* unable to provide informed consent due to cognitive deficit, serious mental illness, or active substance use

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women are eligible to participate
Enrollment: 50 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Participant attrition | From enrollment to end of 12 week intervention
  Measure of participants who withdraw from the behavioral trial in the intervention and the control groups to determine feasibility of enrolling and retaining individuals in the trial. Approximately 15% attrition is expected in a behavioral clinical trial. Higher levels of attrition relate to lower feasibility.
Intervention acceptability: Satisfaction | Mid-point (6-week) assessment and end of intervention assessment (12-week)
  Participant satisfaction with the intervention: Treatment Satisfaction Questionnaire adapted for behavioral treatment. The measure includes 11 items asked on a Likert-type scale from 1=Extremely Dissatisfied to 7=Extremely Satisfied, with 3 items asked on a 1-5 scale. 1 item will be removed that asks about medication side effects. Scores can range from 10 to 64. Higher scores mean higher satisfaction with the treatment/intervention.
Intervention Acceptability: Treatment burden | At 6-week (mid-point intervention) and 12-weeks (end of intervention)
  The Brief Patient Experiences with Treatment and Self Management will be used. The scale includes 32 items total. Most items use a 5-point Likert-type scale from 1=very easy to 5=very difficult. Some items use a 5-point Likert scale (agreement). And some use a Likert-type frequency/intensity measure from 1=not at all to 5=very much. Does not apply=0. Total scores range from 0 to 150. Higher scores mean higher treatment burden.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | Measured at baseline, 6-weeks (mid-point) and 12-weeks (end of intervention)
  Home blood pressure readings taken x3 and averaged.
Daily physical activity: Accelerometer measured | Collected at baseline pre-randomization, and at 12-weeks (end of intervention)
  7-day accelerometer observation of daily physical activity
Self reported physical activity | Collected at baseline, 6 weeks (mid-point), and 12-weeks (post-intervention)
  Time and intensity of physical activity via the International Physical Activity Questionnaire - Short Form (IPAQ-SF) which are then computed to a continuous score of MET (metabolic equivalents)-minutes per week. Computed as follows: Total PA METmin/week=[(3.3*walking minutes*walking days)+(4.0*moderate activity minutes*moderate activity days)+(8.0*vigorous activity minutes*vigorous activity days)]. Higher scores mean greater physical activity.
Physical Activity Self Efficacy | Collected at baseline, 6-weeks (mid-point) and 12-weeks (post-intervention)
  Confidence to engage in regular physical activity will be measured using the Exercise Self Efficacy Scale. A total of 9 items are asked using a scale from 0=not at all confident to 10=completely confident. Scores range from 0-90. Higher scores mean higher self efficacy.
Physical activity enjoyment | Collected at baseline, 6-weeks (mid-point), and 12-weeks (post-intervention)
  Physical activity enjoyment scale will be used. The scale has 18 items and each item is asked on a 1 to 7 scale. Scores may range from 18-126. Higher scores mean higher enjoyment and perceived positive outcomes from exercise/physical activity.
Social support for physical activity | Collected at baseline, 6-weeks (mid-point), and 12-weeks (post-intervention)
  Social support for exercise behaviors scale will be used that includes 10 items asked on a scale from 1=none to 5=very often, there is also an option for does not apply. Scores range from 10-50. Higher scores mean more social support for physical activity.

OTHER OUTCOMES:
General Social Support | Collected at baseline, 6-weeks (mid-point), and 12-weeks (post-intervention)
  Medical outcomes study social support scale will be used to assess global social support. The scale includes 19 items and the overall support index is calculated by taking the mean of all of the items resulting in a range from 1-5. Scores can be transformed to a 0-100 score by the following equation: 100*((observed score-minimum possible score)/(maximum possible score-minimum possible score)). Higher scores mean greater social support.
Health related quality of life | Collected at baseline, 6-weeks (mid-point), and 12-weeks (post-intervention)
  The Short Form Health Survey-12 (SF-12) will be used to assess Health related quality of life (HRQoL) which asks about physical and emotional health in the past 4 weeks using 12 items. In scoring, all items are coded to yield a total score between 0 and 100 such that higher scores mean better HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Kaylee B Crockett, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Department of Family & Community Medicine; University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Pilot trial; Certificate of confidentiality